CLINICAL TRIAL: NCT05101291
Title: Fractional Spinal Anesthesia and Systemic Hemodynamics in Frail Elderly Hip Fracture Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgard, Associate Professor, Head of Department, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Fractional Spinal LidCO
Record Dates: First submitted 2021-10-06; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Hip Fractures; Anesthesia; Hypotension Drug-Induced; Cardiac Output, Low
Keywords: hip fracture; Spinal anaesthesia; fractional; hypotension; cardiac output; elderly patients
MeSH Terms: conditions — Hip Fractures; Hypotension; Cardiac Output, Low | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Single arm, open label investigation on the hemodynamic effect of fractional spinal anaesthesia as measured by lithium dilution cardiac output monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fractional spinal anaesthesia (Experimental): After FIC block or femoral nerve block with ropivacaine 3.5mg/ml 20-40ml. The LiDCOplus was calibrated with 0.3-0.45 mmol lithium based on body weight. After calibration and baseline parameter registration, the LiDCOplus system provided cardiac output variables A dural puncture by a 18G Tuohy needle was performed either between the L2 - L3 or the L3 - L4 interspaces, preferably using a mid-line approach. A catheter 20G was then inserted 4-5 cm into the intrathecal space. A solution (10 ml) of 1.5 mg/ml bupivacaine and 10 µg/ml fentanyl was prepared. Intrathecal anaesthesia was induced by giving 1,5 ml (2.25 mg of bupivacaine and 15 µg of fentanyl) of the solution, followed by a second 1.5 ml injection after 25 min.
  MAP was maintained with a norepinephrine to target a MAP >65mmHg or to avoid a > 30% decline in MAP from baseline. Invasive haemodynamic parameters were recorded every 5 min for 45 min after initial intrathecal dose was given.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — Interventional anaesthesia provided through an indwelling spinal catheter was administered according to protocol
  Other Names: Fractional spinal anaesthesia

SUMMARY:
Aging and frailty make the elderly patients susceptible to hypotension following spinal anaesthesia. The systemic haemodynamic effects of spinal anaesthesia are not well known. In this study, we examine the systemic haemodynamic effects of fractional spinal anaesthesia following intermittent microdosing of a local anesthetic and an opioid.

We included 15 patients aged over 65 with considerable comorbidities, planned for emergency hip fracture repair. Patients received a spinal catheter and cardiac output monitoring using the LiDCOplus system. Invasive mean arterial pressure (MAP), cardiac index, systemic vascular resistance index, heart rate and stroke volume index were registered. Two doses of bupivacaine 2,25 mg and fentanyl 15µg were administered with 25 minutes in between. Hypotension was defined as a fall in MAP by >30% or a MAP <65 mmHg

DETAILED DESCRIPTION:
We daily screened patients planned for hip fracture surgery and these were identified through the theatre planning software (Orbit, TietoEVRY, Espoo, Finland). Nottingham Hip Fracture Score was calculated. This scoring system includes objective factors like age, sex, dementia, previous cancer, living facility and comorbidity. NHFS varies from 1-10 with higher numbers correlated to higher 30-day mortality. ASA grade was also recorded after study inclusion.

After arriving to the preoperative area, patients were given 5 liters of oxygen on a face mask and ECG and pulse-oximetry monitoring were started. Oral premedication with standardized doses of paracetamol and oxycodone was given orally, followed by the placement of a venous 18G cannula in an antecubital vein and a radial arterial catheter (20G). The patient was also given a fascia iliaca compartment (FIC) block, or an ultrasound guided femoral nerve block with ropivacaine 3.5mg/ml 20-40ml, to decrease discomfort when given the neuraxial block. In addition, the LiDCOplus (LiDCO Group Plc, London, England) system was set up according to manufacturer's instructions. The system was calibrated with 0.3-0.45 mmol lithium chloride depending on body weight. After calibration and baseline parameter registration, the LiDCOplus system provided cardiac output variables and based on these and the invasive blood pressure, haemodynamic variables could be derived.

Following aseptic skin preparation of the lumbar area, a subarachnoid puncture by a 18G Tuohy needle was performed either between the L2 - L3 or the L3 - L4 interspaces, preferably using a mid-line approach. An intrathecal catheter 20G was then inserted 4-5 cm into the intrathecal space. This technique of a continues spinal anaesthesia (CSA) was performed on all patients by one physician (FO). A solution (10 ml) containing 1.5 mg/ml bupivacaine and 10 µg/ml fentanyl was prepared. Intrathecal anaesthesia was induced by giving 1,5 ml (2.25 mg of bupivacaine and 15 µg of fentanyl) of the solution, followed by a second 1.5 ml injection after 25 min (i.e., a total intrathecal dos of 4.5 mg of bupivacaine and 30 µg of fentanyl). Sensory level was monitored by "cold spray". Hemodynamic recordings were performed every 5 minutes up until 45 minutes after initial intrathecal dose when research monitoring was terminated. The patient was then operated in the pre-planned time slot and was further managed at the discretion of the attending anesthetist.

ELIGIBILITY:
Inclusion Criteria:

1. patient with hip fracture,
2. >65 years of age,
3. ASA ≥2, 4) scheduled for neuraxial anaesthesia and 5) mentally intact to give informed consent. This could also be given by next-of-kin, if the patient was cognitively impaired.

Exclusion Criteria:

1. lithium or anticoagulation medication,
2. planned for general anaesthesia,
3. ongoing atrial fibrillation,
4. if surgery was delayed >72 hours,
5. lack of informed consent and
6. patient agitation requiring intermittent sedation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | 45 minutes
  Mean arterial pressure change over time and in relation to intrathecal dosing
Cardiac Output | 45 minutes
  Cardiac Output change over time and in relation to intrathecal dosing
Systemic Vascular Resistance Index | 45 minutes
  Systemic vascular resistance indexchange over time and in relation to intrathecal dosing
Elastance | 45 minutes
  Arterial Elastance change over time and in relation to intrathecal dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Nellgård, MD PhD, Study Director — Head of det
Locations (1):
- Sahlgrenska University Hospital /Mölndal, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
The number of participants is low and anonymity would be difficult to guarantee.

REFERENCES:
- [Background] Griffiths R, Babu S, Dixon P, Freeman N, Hurford D, Kelleher E, Moppett I, Ray D, Sahota O, Shields M, White S. Guideline for the management of hip fractures 2020: Guideline by the Association of Anaesthetists. Anaesthesia. 2021 Feb;76(2):225-237. doi: 10.1111/anae.15291. Epub 2020 Dec 2. PMID 33289066
- [Background] Nakasuji M, Suh SH, Nomura M, Nakamura M, Imanaka N, Tanaka M, Nakasuji K. Hypotension from spinal anesthesia in patients aged greater than 80 years is due to a decrease in systemic vascular resistance. J Clin Anesth. 2012 May;24(3):201-6. doi: 10.1016/j.jclinane.2011.07.014. PMID 22537572
- [Background] Jakobsson J, Kalman SH, Lindeberg-Lindvet M, Bartha E. Is postspinal hypotension a sign of impaired cardiac performance in the elderly? An observational mechanistic study. Br J Anaesth. 2017 Dec 1;119(6):1178-1185. doi: 10.1093/bja/aex274. PMID 29040402
- [Background] Wiles MD, Moran CG, Sahota O, Moppett IK. Nottingham Hip Fracture Score as a predictor of one year mortality in patients undergoing surgical repair of fractured neck of femur. Br J Anaesth. 2011 Apr;106(4):501-4. doi: 10.1093/bja/aeq405. Epub 2011 Jan 28. PMID 21278153